CLINICAL TRIAL: NCT06493942
Title: Clinical Evaluation of Bioactive Versus Filled Resin Based Pit & Fissure Sealants in First Permanent Molars: A Randomized Controlled Trial
Brief Title: Clinical Efficiency of Bioactive Pit and Fissure Sealant
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samaa Salah Eldin Abd Elfattah, Assistant lecturer in pediatric dentistry department, faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BPFS
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Pit and Fissure Sealant
Keywords: dental sealant; pit and fissure sealant; fissure sealant; Bioactive dental sealant; Tooth sealant; Fissure sealants; Dental sealants; Pit sealants
MeSH Terms: conditions — Van der Woude syndrome | interventions — Ultra Seal XT

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding to participants : will not know either the intervention or the comparator will be applied to their teeth Blinding to investigator: covering the 2 syringes with opaque seal to avoid performance bias Blinding to outcomes assessor: to overcome detection bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (A) (Active Comparator): Fluoride releasing filled resin based pit and fissure sealant using UltraSeal XT™ plus by Ultradent
  Interventions: Other: UltraSeal XT™ plus by Ultradent
- Interventional group (B) (Experimental): Bioactive pit and fissure sealant using BioCoat® by Premier®
  Interventions: Other: BioCoat® by Premier®

INTERVENTIONS:
Other: BioCoat® by Premier® — BioCoat is a 56% filled resin formula that provides added strength and excellent long-term resistance to wear ؤomparable to flowable composites.
  Arms: Interventional group (B)
Other: UltraSeal XT™ plus by Ultradent — UltraSeal XT plus is a 58%-filled resin fluoride-releasing sealant. It is strong and has high wear resistant
  Arms: Control group (A)

SUMMARY:
This study will compare the performance of newly introduced bioactive resin based pits and fissure sealant versus fluoride releasing filled resin based pits and fissure sealant in posterior molars prone to carious lesions of fissures in patients at risk of caries. Visual tactile examination and VistaCAM will be used for evaluation.

DETAILED DESCRIPTION:
New bioactive resin pits and fissures sealant BioCoat® by Premier® presenting SmartCap™ Technology involving semi-permeable resin microcapsules. The rechargeable SmartCap microcapsules are filled with ionic solutions of fluoride, calcium and phosphate, supposing greater fluoride uptake in the presence of calcium and phosphate ions.

With no enough evidence based information in literature about using bioactive fissure sealants in susceptible fissures , it isd beneficial to evaluate the newly introduced material using a randomized clinical trial to test the null hypothesis that bioactive resin pit and fissure sealant will have the same clinical performance as flouride releasing filled resin based pit and fissure sealant in susceptible fissures.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria of participants:

  * Patients with caries susceptible fiss- ures in fully erupted first permanent molars showing nosigns of caries.
  * Co-operative patients approving to part- icipate in the trial.
  * Good oral hygiene.
* Inclusion Criteria of teeth:

  * Caries susceptible occlusal pits and fissures.
  * Intact contact with opposing teeth.
  * Teeth with no previous restorations in other surfaces.

Exclusion Criteria:

* Exclusion criteria of participants:

  * patients with Disabilities, systemic disease or severe medical complications.
  * patients have allergic history concerning methacrylate.
  * patients with rampant caries, xerostomia, evidence of severe bruxism, clenching, or tempromandibular joint disorders
  * participants who show lack of compliance.
* Exclusion criteria of teeth:

  * Carious pits and fissures.
  * Developmental tooth defect.
  * Partially erupted teeth
  * Periapical pathology or signs of pulpal pathology.
  * Tooth hypersensitivity.
  * Heavy occlusion and occlusal contacts.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Retention of sealant | 1 year
  rate of sealant loss

SECONDARY OUTCOMES:
Caries incidence | 1 year
  Rate of caries progression

IPD SHARING:
Plan to Share IPD: Undecided